CLINICAL TRIAL: NCT04038242
Title: A Resilience Promotion Program for Parents of Children With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: UW 19-436
Record Dates: First submitted 2019-07-17; First posted 2019-07-30 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Parents of Children With Cancer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resilience promotion program (Experimental): Subjects in the intervention group will participate in an eight-session resilience promotion program.
  Interventions: Other: Resilience promotion program
- Treatment as usual (No Intervention): Treatment as usual for subjects in the control group.

INTERVENTIONS:
Other: Resilience promotion program — Resilience Promotion Program consists of eight sessions. Except the first orientation session and the last review session, other six sessions focus on cultivating the five internal resiliency factors (physical, behavioral, cognitive, emotional and spiritual). There are two sessions for behavioral factor, including one special to deal with the relationships between parents and children.
  Arms: Resilience promotion program

SUMMARY:
Cancer is a leading cause of death for children. With the increasing incidence of childhood cancer, the mental health problems emerge in those parents struggle with their children's life-threatened disease. Caring for children with cancer is described as life-changing experience and overwhelming stress for parents. Many studies have been conducted to screen the psychological distress for these parents and found a considerable percentage of them suffering from depressive symptoms. Poorer quality of life was also found in parents of children with cancer when compared to parents of children without cancer. Additionally, parental distress interacted with children's emotions and could have detrimental effects on children's both physical and mental health. Therefore, it is important to take measures improving the mental health for parents of children with cancer.

Although current various psychological interventions illustrated small to moderate improvements of mental health for parents of children with cancer, the total effect base on a systematic review was not statistically significant. The purpose of these interventions was predominantly to treat negative mental health problems such as depression and no recognized effective psychological interventions were available for parents of children with cancer until now. Along with the paradigm shift from problem-oriented approach to nurturing strengths in the post-modern period, instead of exclusively treating mental health problems, researchers payed more attention to positive therapy such as resilience promotion program. Resilience usually refers to the ability to adapt adverse conditions and maintain positive status. Resilience studies are mounting since the flourishing of positive psychology movement and meaningful results were gained from corresponding intervention program concentrating on resilience promotion in adolescent education, handling chronic disease and recovery of breast cancer. However, there is a lack of targeted resilience promotion program for parents of children with cancer. The results of our pilot study showed low levels of resilience in parents of children with cancer and strong associations among parental resilience, quality of life and depression. It indicates that the increase in resilience can benefit for the mental health of parents. Therefore, a resilience promotion program will be conducted to examine efficacy for parents of children with cancer.

ELIGIBILITY:
Inclusion Criteria:

* having a child (0-19 years old) with cancer diagnosis.
* Chinese resident and able to read Chinese and speak Mandarin.

Exclusion Criteria:

* having physical impairment or cognitive and learning problems identified from family history of medical records.
* attending other researches.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2019-08-13 (Actual); Primary Completion 2020-07-21 (Actual); Study Completion 2020-07-21 (Actual)

PRIMARY OUTCOMES:
Change in levels of resilience from baseline to 6-month follow-up between intervention and control group | 6-month follow-up
  The primary outcome measure is the resilience of subjects at 6-month follow-up when compare to baseline. The Connor-Davison resilience scale will be used to assess participants' resilience. The total score ranges from 0-100 and higher score reflecting higher levels of resilience.

SECONDARY OUTCOMES:
Levels of resilience at baseline | baseline
  The Connor-Davison resilience scale will be used to assess participants' resilience. The total score ranges from 0-100 and higher score reflecting higher levels of resilience.
Change in levels of resilience from baseline to 2-month follow-up between intervention and control group | 2-month follow-up
  The Connor-Davison resilience scale will be used to assess participants' resilience. The total score ranges from 0-100 and higher score reflecting higher levels of resilience.
Levels of quality of life at baseline | baseline
  The Short Form of Medical Outcomes will be used to measure quality of life. The total score ranges from 0.32 for the worst health state to 1 for full health.
Change in levels of quality of life from baseline to 2-month follow-up between intervention and control group | 2-month follow-up
  The Short Form of Medical Outcomes will be used to measure quality of life. The total score ranges from 0.32 for the worst health state to 1 for full health.
Change in levels of quality of life from baseline to 6-month follow-up between intervention and control group | 6-month follow-up
  The Short Form of Medical Outcomes will be used to measure quality of life. The total score ranges from 0.32 for the worst health state to 1 for full health.
Levels of depression at baseline | baseline
  Self-rating depression scale will be used to measure depression. The total score ranges from 20 to 80. Higher total score indicates more serious depression status.
Change in levels of depression from baseline to 2-month follow-up between intervention and control group | 2-month follow-up
  Self-rating depression scale will be used to measure depression. The total score ranges from 20 to 80. Higher total score indicates more serious depression status.
Change in levels of depression from baseline to 6-month follow-up between intervention and control group | 6-month follow-up
  Self-rating depression scale will be used to measure depression. The total score ranges from 20 to 80. Higher total score indicates more serious depression status.
Levels of anxiety at baseline | baseline
  Self-rating anxiety scale will be used to measure anxiety. The total score ranges from 25 to 100 and higher score reflects worse anxiety status.
Change in levels of anxiety from baseline to 2-month follow-up between intervention and control group | 2-month follow-up
  Self-rating anxiety scale will be used to measure anxiety. The total score ranges from 25 to 100 and higher score reflects worse anxiety status.
Change in levels of anxiety from baseline to 6-month follow-up between intervention and control group | 6-month follow-up
  Self-rating anxiety scale will be used to measure anxiety. The total score ranges from 25 to 100 and higher score reflects worse anxiety status.
Levels of stress at baseline | baseline
  The perceived stress scale will be used to measure stress. The total score ranges from 0 to 40. Higher total score suggests more perceived stress.
Change in levels of stress from baseline to 2-month follow-up between intervention and control group | 2-month follow-up
  The perceived stress scale will be used to measure stress. The total score ranges from 0 to 40. Higher total score suggests more perceived stress.
Change in levels of stress from baseline to 6-month follow-up between intervention and control group | 6-month follow-up
  The perceived stress scale will be used to measure stress. The total score ranges from 0 to 40. Higher total score suggests more perceived stress.

CONTACTS AND LOCATIONS:
Overall Officials: Yuan Hui Luo, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- University of Hong Kong, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Luo Y, Li HCW, Cheung AT, Ho LLK, Xia W, Zhang J. Evaluating the experiences of parents of children with cancer engaging in a mobile device-based resilience training programme: a qualitative study. Support Care Cancer. 2022 Jul;30(7):6205-6214. doi: 10.1007/s00520-022-07066-7. Epub 2022 Apr 20. PMID 35441899
- [Derived] Luo Y, Xia W, Cheung AT, Ho LLK, Zhang J, Xie J, Xiao P, Li HCW. Effectiveness of a Mobile Device-Based Resilience Training Program in Reducing Depressive Symptoms and Enhancing Resilience and Quality of Life in Parents of Children With Cancer: Randomized Controlled Trial. J Med Internet Res. 2021 Nov 29;23(11):e27639. doi: 10.2196/27639. PMID 34847060